CLINICAL TRIAL: NCT00022139
Title: A Phase II Trial of Preoperative Radiation and Chemotherapy (Paclitaxel, Carboplatin, and Continuous Infusion 5-FU) for Locally Advanced Esophageal Cancer
Brief Title: Radiation Therapy and Paclitaxel, Carboplatin, and Fluorouracil Followed by Esophagectomy in Treating Patients With Locally Advanced Cancer of the Esophagus or Gastroesophageal Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0044; NCI-2012-02394 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000068789 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-08-10; First posted 2003-03-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage III gastric cancer; stage II esophageal cancer; stage III esophageal cancer; adenocarcinoma of the stomach; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Carboplatin; Fluorouracil; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- carboplatin + paclitaxel + fluorouracil + radiation + surgery (Experimental): Patients receive carboplatin IV and paclitaxel IV over 3 hours on days 1 and 22 and fluorouracil IV continuously on days 1-42. Beginning on day 1 of chemotherapy, patients undergo radiotherapy to the esophagus 5 days a week for 5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease at 4-8 weeks after completion of radiotherapy undergo esophagectomy and complete dissection of the mediastinal and perigastric lymph nodes. Beginning 8 weeks after surgery, patients who underwent curative resection may receive a maximum of 2 additional courses of paclitaxel and carboplatin in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed at baseline, before chemotherapy on days 1 and 22, and within 2 weeks before surgery.
  Patients are followed every 3 months for 4 years.
  Interventions: Drug: carboplatin; Drug: fluorouracil; Drug: paclitaxel; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin
Drug: fluorouracil
Drug: paclitaxel
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy, such as paclitaxel, carboplatin, and fluorouracil, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving radiation therapy with chemotherapy and giving them before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: This phase II trial is studying how well giving radiation therapy together with combination chemotherapy followed by esophagectomy works in treating patients with locally advanced cancer of the esophagus or gastroesophageal junction.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pathologic complete response rate in patients with locally advanced cancer of the esophagus or gastroesophageal junction treated with radiotherapy administered concurrently with paclitaxel, carboplatin, and fluorouracil before esophagectomy.
* Determine the tolerability of this regimen in these patients.
* Determine the tumor response rate in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Assess the relationship between the presence of genetic polymorphisms in these patients and the toxicity of this regimen.

OUTLINE: This is a multicenter study.

Patients receive carboplatin IV and paclitaxel IV over 3 hours on days 1 and 22 and fluorouracil IV continuously on days 1-42. Beginning on day 1 of chemotherapy, patients undergo radiotherapy to the esophagus 5 days a week for 5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease at 4-8 weeks after completion of radiotherapy undergo esophagectomy and complete dissection of the mediastinal and perigastric lymph nodes. Beginning 8 weeks after surgery, patients who underwent curative resection may receive a maximum of 2 additional courses of paclitaxel and carboplatin in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before chemotherapy on days 1 and 22, and within 2 weeks before surgery.

Patients are followed every 3 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma or adenocarcinoma of the thoracic esophagus (below 20 cm) or gastroesophageal junction

  * Surgically resectable disease (T1-3; NX, N0, or N1; M1a)
  * T4 tumors that are not unequivocally unresectable allowed
  * Celiac lymph node (stations 15-20) involvement allowed
* Must be considered a potential surgical candidate by a thoracic or general surgeon
* No supraclavicular lymph node involvement by palpation, biopsy, or radiograph (greater than 1.5 cm)
* No distant metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

  * Patients with ECOG 2 must be considered good candidates for study by treating oncologists

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 3 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No New York Heart Association class III or IV heart disease

Other

* No uncontrolled infection
* No other severe underlying disease that would preclude study participation
* No grade 2 or greater peripheral neuropathy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for esophageal cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to anticipated fields of study radiotherapy

Surgery

* Not specified

Other

* No concurrent diuretics
* No concurrent amifostine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2002-01; Primary Completion 2005-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Proportion of successes | Up to 4 years

SECONDARY OUTCOMES:
Toxicity-free rate | Up to 4 years
Clinical tumor response | Up to 4 years
Pathologic tumor response | Up to 4 years
Time to disease progression | Up to 4 years
Surgical outcome | Up to 4 years
Survival | Up to 4 years
Time to treatment failure | Up to 4 years
Quality of life | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (35):
- United States (35):
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota

REFERENCES:
- [Background] Jatoi A. Aggressive multimodality therapy for patients with locally advanced esophageal cancer: is there a role for amifostine? Semin Oncol. 2003 Dec;30(6 Suppl 18):72-5. doi: 10.1053/j.seminoncol.2003.11.013. PMID 14727244
- [Result] Jatoi A, Martenson JA, Foster NR, McLeod HL, Lair BS, Nichols F, Tschetter LK, Moore DF Jr, Fitch TR, Alberts SR; North Central Cancer Treatment Group (N0044). Paclitaxel, carboplatin, 5-fluorouracil, and radiation for locally advanced esophageal cancer: phase II results of preliminary pharmacologic and molecular efforts to mitigate toxicity and predict outcomes: North Central Cancer Treatment Group (N0044). Am J Clin Oncol. 2007 Oct;30(5):507-13. doi: 10.1097/COC.0b013e31805c139a. PMID 17921712
- [Result] Jatoi A, Martenson J, Mahoney MR, Lair BS, Brindle JS, Nichols F, Caron N, Rowland K, Tschetter L, Alberts S. Results of a planned interim toxicity analysis with trimodality therapy, including carboplatin AUC = 4, paclitaxel, 5-fluorouracil, amifostine, and radiation for locally advanced esophageal cancer: preliminary analyses and treatment recommendations from the North Central Cancer Treatment Group. Int Semin Surg Oncol. 2004 Nov 8;1(1):9. doi: 10.1186/1477-7800-1-9. PMID 15533252